CLINICAL TRIAL: NCT05356572
Title: A Single-center, Open, Randomized, Non-controlled, Comparative Pre-market Investigation to Evaluate the Performance of a Skin Preparation Device for Removal of Hyperkeratotic Skin
Brief Title: A Pre-market Study to Evaluate the Performance and Safety of a Skin Preparation Device for Removal of Dry Crusty Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mirka Ltd (Industry)
Collaborators: Clinius Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCIREP2204
Record Dates: First submitted 2022-04-14; First posted 2022-05-02 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Keratosis, Actinic; Actinic Lesion; Solar Keratosis/Sunburn; Hyperkeratosis; Hyperkeratotic Callus; Hyperkeratotic; Lesion; Hyperkeratotic Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic; Sunburn; Keratoderma, Palmoplantar, Epidermolytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Skin Preparation Device versus Disposable Dermal Curette (Active Comparator)
  Interventions: Device: Investigational Skin Preparation Device; Device: UMDNS 13-230 / Biopsy punch (Dermal Curette)
- Investigational Skin Preparation Device versus Abrasive Pad for Skin Preparation (Active Comparator)
  Interventions: Device: Investigational Skin Preparation Device; Device: GMDN 47102 / Electrode Skin Abrasive Pad

INTERVENTIONS:
Device: Investigational Skin Preparation Device — Removal of hyperkeratotic skin with Investigational Skin Preparation Device
Device: GMDN 47102 / Electrode Skin Abrasive Pad — Removal of hyperkeratotic skin with Abrasive Pad for Skin Preparation
  Arms: Investigational Skin Preparation Device versus Abrasive Pad for Skin Preparation
Device: UMDNS 13-230 / Biopsy punch (Dermal Curette) — Removal of hyperkeratotic skin with Disposable Dermal Curette
  Arms: Investigational Skin Preparation Device versus Disposable Dermal Curette

SUMMARY:
In this clinical one-site investigation the performance and safety of a skin preparation device will be evaluated for removing hyperkeratotic skin prior to further medical treatment. Comfort and pain during skin preparation, as well as performance and safety of device, will be compared to comparators on separate skin areas for every subject.

ELIGIBILITY:
Inclusion Criteria:

* Attending the clinic for treatment of actinic keratosis using daylight photodynamic therapy
* Age: 18 - 100 years.
* Available for two follow-up visits: two weeks after treatment and 4 months after treatment
* Provision of informed consent i.e., subject must be able to understand and sign the patient Information and Consent Form
* Subject have been informed on the nature, the scope and the relevance of the study

Exclusion Criteria:

* Known or suspected allergy/hypersensitivity to phenol formaldehyde
* Wound at the skin site to be treated
* Documented skin disease at the time of enrollment, as judged by the investigator
* Previously enrolled in the present investigation
* Inclusion in other ongoing investigations simultaneously that would preclude the subject from participating in this investigation as judged by the investigator
* Actinic keratosis treatment obtained within last 6 months
* Involvement in the planning and conduct of the clinical investigation (applies to all investigation site staff and third party vendor)
* Any subject that according to Medical Research Act, paragraphs 7-10, is deemed unsuitable for study enrolment.
* Complications that would increase wound risks if investigational product would be used.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

PRIMARY OUTCOMES:
Grade of hyperkeratotic skin removal | Day 0
  Sufficient hyperkeratotic skin removal in comparison to comparative methods. The removal of hyperkeratotic skin is assessed visually and by palpation.
  Removal of hyperkeratotic skin measurement grades: All hyperkeratotic skin removed, Partial hyperkeratotic skin removed, None hyperkeratotic skin removed.

SECONDARY OUTCOMES:
Grade of injury to skin / grade of skin irritation / grade of allergic skin reaction | Day 0
  Investigator assessment of adverse effects on skin in comparison to the comparative methods.
  Grade of injury to skin: none, mild, moderate, severe. Grade of skin irritation: none, mild, moderate, severe. Grade of allergic skin reaction: none, mild, moderate, severe.
Grade of skin irritation / grade of allergic skin reaction | 14 day follow-up
  Investigator assessment of adverse effects on skin in comparison to the comparative methods.
  Grade of skin irritation: none, mild, moderate, severe. Grade of allergic skin reaction: none, mild, moderate, severe.
Duration of operation time per treated skin area | Day 0
  Operation time assessed by the mean difference in time per treated skin area to remove the hyperkeratotic skin in comparison to comparative methods.
Presence of actinic keratosis | Day 0
  Presence of actinic keratosis (AK) is measured by number of different grades of AK lesions.
  Number of different grades of AK lesions: None, Grade I AK lesions, Grade II AK lesions, Grade III AK lesions.
Clearance of actinic keratosis | 4th month follow-up
  Number of different grades of actinic keratosis (AK) lesions are measured: None, Grade I AK lesions, Grade II AK lesions, Grade III AK lesions.
  Actinic keratosis clearance is assessed as the number of cleared actinic keratosis lesions at 4th month follow-up divided by the actinic keratosis lesion number at Day 0. Clearance will be reported in %. A high %-value means a high number of cleared lesions.
Physician comfort during skin preparation using an investigator questionnaire | Day 0
  Rate of physician comfort when comparing the investigational product versus comparative methods. The endpoint will utilize a questionnaire for the investigator/nurse to fill in.
Subject comfort during skin preparation using a subject questionnaire | Day 0
  Rate of subject comfort (including skin sensation and heating of skin) when comparing the investigational product with comparative methods. The endpoint will utilize a questionnaire for the subject to fill in.
  Skin sensation during skin preparation: Very pleasant, Pleasant, Neutral, Unpleasant, Very unpleasant.
  Heating of skin during skin preparation: None, Mild temperature rise, Moderate temperature rise, High temperature rise, Burning.
Subject pain sensation during skin preparation | Day 0
  Rate of pain using visual analogue scale (VAS). VAS: 0 - 10 (0= No pain and 10 = worst possible pain)
Subject pain sensation during daylight photodynamic treatment | Day 0
  Rate of pain using visual analogue scale (VAS). VAS: 0 - 10 (0= No pain and 10 = worst possible pain)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna H Hagman, M.D, PhD, Principal Investigator — Vaasa Central Hospital, Vaasa, Finland
Locations (1):
- Vaasa Central Hospital, Vaasa, Finland

IPD SHARING:
Plan to Share IPD: No